CLINICAL TRIAL: NCT05117203
Title: Immediate Effects of Dynamic Electrostimulation on the Abdominal Muscles in Healthy Individuals, Assessed by Ultrasound: an Experimental Study
Brief Title: Dynamic Electrostimulation on the Abdominal Muscles in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Lorena Álvarez del Barrio, Principal Investigator, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ETICA-ULE-009-2020
Record Dates: First submitted 2021-10-25; First posted 2021-11-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: Whole body electrostimulation; healthy; abdominal muscles; ultrasound; RUSI; WB-EMS
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WB-EMS group (Experimental)
  Interventions: Device: WB-EMS (Whole body electrostimulation)
- EMS group (Experimental)
  Interventions: Device: EMS
- Control group (Sham Comparator)
  Interventions: Device: WB-EMS off

INTERVENTIONS:
Device: WB-EMS (Whole body electrostimulation) — Application of physical exercise and electrical stimulation on the abdominal muscles through the WB-EMS during 20 minutes training session with specific exercise (CORE)
  Arms: WB-EMS group
Device: EMS — Application of physical exercise and electrical stimulation on the abdominal muscles through the EMS during 20 minutes training session with specific exercise (CORE)
  Arms: EMS group
Device: WB-EMS off — Application of physical exercise without electrical stimulation on the abdominal muscles through the WB-EMS off during a 20 minutes training session with specific exercise (CORE).
  Other Names: Control group
  Arms: Control group

SUMMARY:
To determine the immediate effects on the abdominal musculature, assessed by ultrasound (RUSI), due to the application of electrostimulation using whole body electrostimulation together with physical exercise in healthy people and to compare with the application of local EMS in the abdominal area and the same physical exercise session. The same intervention is carried out for the control group as the WB-EMS group but simulated.

DETAILED DESCRIPTION:
Evaluation of the immediate changes in the thickness of the abdominal muscles (Transversus abdominis, Internal and External Oblique and Rectus abdominis) and in the Interrectus distance after the physical exercise session together with whole body electrostimulation or local electrostimulation assessed by ultrasound (RUSI) in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Good medical history without injury or chest pain in the past year
* No surgeries in the previous year.

Exclusion Criteria:

* Upper body mass index 30 Kg/m2
* Level of professional or elite sports activity
* Hyperventilation / hypercapnia and score above 23 points on the Nijmegen questionnaire
* Present any contraindication regarding the WB-EMS/EMS
* Viral o bacterial infections
* Arterial circulatory disorders, advanced arteriosclerosis
* Women during their menstrual period
* Type I diabetes, hemophilia, bruises, bleeding, cognitive deficit, fibromyalgia, congenital diseases with muscle-skeletal alterations at the level of the back and lower extremities, scoliosis, protrusion or disc herniation, medication consumption, abdominal surgeries (scars or keloids), abdominal muscle injury.
* Presence of chronic low back, hip or thigh pain

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Measurement of muscle thickness of the abdominal muscles by ultrasound through the technique "Rehabilitative Ultrasound Imaging" (RUSI). | One day
  Measure muscle thickness before and after exercise with electrostimulation
Measurement of the Distance between Rectus abdominis using ultrasound (RUSI) | One day
  Measure the distance between Rectus abdominis before and after exercise with electrostimulation

SECONDARY OUTCOMES:
International physical activity questionnaire (IPAQ) | One day
  Classification according to low, moderate or high physical activity level
Nijgemen questionnaire | One day
  A level of respiratory distress equal to or higher than 23 points is an exclusion criterion for exclusion from the study
Body height | One day
  Body height in meters
Body weight | One day
  Body weight in kilograms
Body mass index | One day
  Calculation of body mass index in Kg/m2 according to Queletet method
Heart frequency | One day
  Measurement of the heart rate (beats per minute)
Blood pressure | One day
  Measurement of systolic and diastolic blood pressure using a sphygmomanometer
body temperature | one day
  Measurement of body temperature in Celsius with a digital thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de León, Ponferrada, León, Spain